CLINICAL TRIAL: NCT02973737
Title: Pyrotinib Plus Capecitabine Versus Placebo Plus Capecitabine in Patients With HER2+ Metastatic Breast Cancer:a Randomised, Double-blind, Multicentre, Phase 3 Trial
Brief Title: A Study of Pyrotinib Plus Capecitabine in Patients With HER2+ Metastatic Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-BLTN-Ⅲ-MBC-A
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: HER2 Positive Metastatic Breast Cancer
MeSH Terms: interventions — pyrotinib; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm 1 (Experimental): pyrotinib plus capecitabine pyrotinib(400 mg once daily) + capecitabine (2000 mg/m^2 daily, 1000 mg/m^2 BID)
  Interventions: Drug: pyrotinib; Drug: Capecitabine
- arm 2 (Active Comparator): placebo plus capecitabine placebo(400 mg once daily) + capecitabine (2000 mg/m^2 daily, 1000 mg/m^2 BID)
  Interventions: Drug: placebo; Drug: Capecitabine

INTERVENTIONS:
Drug: pyrotinib — 400 mg once daily
  Arms: arm 1
Drug: placebo — 400 mg once daily
  Arms: arm 2
Drug: Capecitabine — 1000 mg/m2 per day on day 1 through 14, every 21 days.

SUMMARY:
Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. This study is a randomized, multi-center, multinational, double blind, active-controlled, parallel design study of the combination of pyrotinib in combination with capecitabine versus placebo plus capecitabine in HER2+ MBC patients, who have prior received anthracyclin, taxane and trastuzumab.

Patients will be randomized in a 2:1 ratio to one of the following treatment arms:

Arm A: pyrotinib (400 mg once daily) + capecitabine (1000 mg/m^2 twice daily) Arm B: placebo (400 mg once daily) + capecitabine (1000 mg/m^2 twice daily) Patients will receive either arm of therapy until the occurrence of death, disease progression, unacceptable toxicity, or other specified withdrawal criterion.

Patients in control group can be provide pyrotinib treatment when they progressed after the placebo plus capecitabine treatment.

DETAILED DESCRIPTION:
This study is a phase 3, randomized, multi-center, multinational, double blind, active-controlled, parallel design study of the combination of pyrotinib in combination with capecitabine versus placebo plus capecitabine in HER2+ MBC patients, who have prior received anthracyclin, taxane and trastuzumab.

Patients will be randomized in a 2:1 ratio to one of the following treatment arms:

Arm A: pyrotinib (400 mg once daily) + capecitabine (1000 mg/m^2 twice daily) Arm B: placebo (400 mg once daily) + capecitabine (1000 mg/m^2 twice daily) Patients will receive either arm of therapy until the occurrence of death, disease progression, unacceptable toxicity, or other specified withdrawal criterion.

Efficacy assessments will be performed at screening, every 6 weeks until cycle 18, every 12 weeks thereafter.

Patients in control group can be provide pyrotinib treatment when they progressed after the placebo plus capecitabine treatment. Pyrotinb will be administrated until the patients reached progress again or wit

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 and ≤75 years.
2. ECOG performance status of 0 to 1.
3. Life expectancy of more than 12 weeks.
4. According to RECIST 1.1, at least one measurable lesion exists
5. Histologically or cytologic confirmed HER2 positive advanced breast cancer which failed prior therapies.
6. Prior treatment with trastuzumab(≥2 cycles in the metastatic setting, or ≥3 months in adjuvant setting), and the patients are not available for the trastuzumab or lapatinib
7. Previously reveived both Anthracyclin and Taxane.
8. Required laboratory values including following parameters:

   ANC: ≥ 1.5 x 10^9/L; Platelet count: ≥ 90 x 10^9/L; Hemoglobin: ≥ 9.0 g/dL; Total bilirubin: ≤ 1.5 x upper limit of normal (ULN); ALT and AST: ≤ 2 x ULN(patients with liver metastases: </= 5 x ULN); BUN and Creatinine: ≤ 1.5 x ULN;LVEF: ≥ 50%;QTcF: < 470 ms.
9. Signed informed consent

Exclusion Criteria:

1. Received previous therapy with lapatinib, neratinib, pyrotinib or any other HER2 directe tyrosine kinase inhibitor.
2. Received previous therapy with capecitabine.
3. History of receiving chemotherapy, target-therapy or investigational treatment within 28 days prior to randomization. Received hormone therapy within 7 days prior to randomization.
4. Brain metastases that are untreated, symptomatic, or require therapy to control symptoms.
5. Current severe, uncontrolled systemic disease.
6. Unable or unwilling to swallow tablets.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Estimated 10 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Estimated 10 months
Safety(adverse Events [AEs] and Serious Adverse Events [SAEs]) | From infromed consent through 28 days following treatment completion
Duration of Response (DOR) | Estimated 10 months
Clinical Benefit rate (CBR) | Estimated 10 months
Overall Survival (OS) | Estimated 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- 307 Hospital Affiliated to Academy Military Medical Science, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes